CLINICAL TRIAL: NCT02857699
Title: Prospective Observational Study to Investigate the Added Value of the Health Related Quality of Life and Patient Reported Symptoms in the Identification of the Recommended Phase II Dose in Phase I Trials of Molecularly Targeted Therapies.
Acronym: QoL Phase I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Collaborators: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2013-07
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Solid Tumors; Quality of Life
Keywords: Quality of life; Phase I trials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective cohort of 250 patients with solid tumours included in phase I clinical trials of targeted agents will be enrolled. Patients will be treated with MTA in mono therapy or in association with chemotherapy or other targeted agents in 4 large phase I centers.

Patients from trials investigating chemotherapy alone will not be included. Quality of life will be assessed during the treatment period.

DETAILED DESCRIPTION:
The main objective of phase I dose finding studies is to identify the recommended phase II dose. The primary endpoint is the dose limiting toxicity (DLT) which is generally measured using the NCI common toxicity criteria (NCI-CTCAE) graded scale. This scale, developed for the investigation of cytotoxic chemotherapy administered in a limited number of cycles including rest period, is well adapted to identify the drug effect on organ dysfunction and life threatening events. However it may be less relevant to reflect the patient's feeling regarding the tolerability of the treatment under study resulting in over or under estimation of these toxicities.

Moreover, targeted therapies and more specifically the ones administered orally are given over long periods often with continuous schedules. Moderate toxic side effects lasting over a long period are usually not considered as DLT. The health related quality of life of patients as well as other patient reported outcome including symptom scale in addition to usual NCI CTCAE scale could be a relevant variable to detect intolerable treatments. It has not been studied prospectively to date in phase I trials.

A prospective cohort of 250 patients with solid tumours included in phase I clinical trials of targeted agents will be enrolled. Patients will be treated with MTA in mono therapy or in association with chemotherapy or other targeted agents in 4 large phase I centers.

Patients from trials investigating chemotherapy alone will not be included.

Patients included in a phase I trial will be requested to fill in

* a questionnaire of health related quality of life (the EORTC PAL 15 questionnaire)
* a questionnaire of symptoms (MDASI)
* a questionnaire on symptoms specific of MTA at baseline and at each cycle of treatment and 6 weeks after the end of treatment.

The sponsor of the therapeutic phase I trials will be informed that the present research is running and that it will not interfere with their investigational protocol. Each phase I center has the latitude to propose or not the health-related quality of life research to patients included in a given phase I trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory solid tumor.
* Patient included in a dose finding phase I trial investigating at least one molecularly targeted agent as defined as anticancer agents that selectively target molecular pathways (including monoclonal antibodies) as opposed to DNA, tubulin or cell division machinery will be eligible.
* Phase I/II clinical trials with a dose finding component are also eligible. Trials investigating combinations of MTA with one or several cytotoxic agent(s) are eligible, as well as combinations of MTAs.

Exclusion Criteria:

- Patients with malignant hematologic disease will not be eligible.

Patients included in the following types of phase I trials are not eligible:

* Trials investigating hormonal therapy and biological therapeutics such as immunotherapy, gene therapy and vaccines alone or in combination;
* Trials of cytotoxic agents only;
* Trials investigating radiochemotherapy alone or in combination with chemotherapy or MTA
* Trials whose objectives do not include dose-finding. This includes pharmacokinetic only trials, bioequivalence trials, feasibility trials etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with refractory solid tumor included in a dose finding phase I trial investigating at least one molecularly targeted agent.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association between HR QoL, patient reported symptoms and DLT. | up to six months
  To evaluate whether some toxic side events that are non dose limiting according to the phase I protocol are reported as intolerable by the patients using either specific HR QoL questionnaires or patient reported scales of symptoms
Patient interviews : qualitative comparison versus EORTC PAL 15 questionary | Up to six months
  Identify if some dimensions of the quality of life affected by the treatment are not captured by the EORTC PAL 15 questionaries.
  Interviews will be realized on a sub sample of patients. An explorative qualitative research could evaluate patients' experience of the impact, burden, tolerability or acceptability of phase I anti-cancer drug trials addressing patients' perception of symptoms, functioning and overall quality of life. Interviews results contrasted with the PAL15 questionnaires will enable to determine whether a QoL questionnaire dedicated to phase I trials is necessary and what are the main components felt essential to the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PAOLETTI, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Centre Georges Francois Leclerc, Dijon
  - Institut Curie, Paris
  - Centre Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No